CLINICAL TRIAL: NCT01295866
Title: Evaluation Effects of Nasal Nitric Oxide Measurements Are Associated With Atopy Status in Chronic Nasal Inflammation
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Demin Han, Beijing Tongren Hospital
Other Study IDs: 1129
Record Dates: First submitted 2011-02-11; First posted 2011-02-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-01

CONDITIONS: Hypersensitivity; Rhinitis; Respiratory Tract Diseases; Nasal Polyps; Nitric Oxide
Keywords: chronic nasal inflammation; nasal nitric oxide; atopy
MeSH Terms: conditions — Hypersensitivity; Rhinitis; Respiratory Tract Diseases; Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- nasal nitric oxide, atypy status
  Interventions: Device: nasal nitric oxide

INTERVENTIONS:
Device: nasal nitric oxide

SUMMARY:
Nitric oxide (NO) was considered as a mediator of nasal inflammation and the measurement of nasal nitric oxide (nNO) may assist in the diagnosis of nasal inflammation. Few data exists comparing nNO with established, larger accepted reference standard for chronic rhinosinusitis (CRS) diagnosis. Moreover, the role of atopic status on nNO in nasal inflammatory diseases has not been reported. The aim of our study was to determine the value of nNO in patients with chronic nasal inflammation, and to assess the relationship between nNO and atopic status in these patients. A total of 131 randomized patients suffering form chronic nonallergic nasal inflammation and 20 healthy volunteers were finally recruited. nNO was measured by NIOX devices. Sinus computed tomography (CT) scan, nasal endoscope and nasal symptoms evaluation were used in the different diagnosis of chronic rhinitis (CR), CRS without nasal polyps (CRSsNP) and CRS with nasal polyps (CRSwNP). Atopic status was confirmed by skin prick test and serum IgE levels. Blood eosinophils were evaluated simultaneously. Relationships among nNO, various atopic characteristics and chronic nasal inflammation were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as CR, CRSsNP or CRSwNP based on the criteria of the European position paper.
* Had at least two or more symptoms, one of which was either nasal blockage/obstruction/congestion or nasal discharge (anterior/posterior nasal drip), and/or facial pain/pressure, and/or reduction or loss of smell;
* Either endoscopic signs of polyps and/or mucopurulent discharge primarily from the middle meatus and/or oedema/mucosal obstruction primarily in the middle meatus.

Exclusion Criteria:

* Pregnancy, lactation, significant psychologic problems, inability to comply with study protocol, children under 18 years of age, systemic diseases affecting the nose (e.g., Wegener's granulomatosis, sarcoid, and acute upper or lower respiratory tract infections within 2 weeks before the inclusion visit)
* Use of systemic corticosteroids within 2 weeks before the inclusion visit, systemic diseases preventing participation in the study, and medical or surgical treatments influencing the study.
* Patients with diagnosed atopic dermatitis and atopic asthma.
* Patients with diagnosed allergic rhinitis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients were prospectively recruited from the Rhinology Clinics of the Otolaryngology, Head and Neck Surgery Department of Beijing TongRen Hospital from January 2010 to November 2010. After application of the exclusion criteria, the study was discussed with 410 consecutive patients with a primary diagnosis of chronic nonallergic nasal inflammation. Of these, 214 agreed to take part in, of which 83 were excluded (57 diagnosed as other nasal diseases such as fungal sinusitis, inverted papilloma and so on, 20 with obviously medicine history in the latest two weeks, and 6 refused to continue). Thus, 131 patients were randomized for inclusion and 20 normal adults were recruited as well in our study.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)